CLINICAL TRIAL: NCT02838043
Title: The Efficacy, Safety, and Tolerability of Probiotics on the Mood and Cognition of Depressed Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Lallemand Health Solutions (Industry); McMaster University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Psychiatrist, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6016312
Record Dates: First submitted 2016-06-02; First posted 2016-07-20 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Major Depressive Disorder; Depression; Depressive Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Depression

ARMS (1):
- Participant (Experimental): All participants will be experimental and receive Probio'Stick.
  Interventions: Dietary Supplement: Probio'Stick

INTERVENTIONS:
Dietary Supplement: Probio'Stick — A combination of the probiotic strains Lactobacillus helveticus and Bifidobacterium longum

SUMMARY:
This study will be an 8-week open-label pilot study examining subjective and objective changes in mood, anxiety, cognition, and sleep before and after the introduction of a probiotic supplement containing Lactobacillus helveticus and Bifidobacterium longum in 10 treatment-naïve participants diagnosed with major depressive disorder (MDD). In order to examine the full composition of the micro biome, the investigators will also be collecting and analyzing fecal samples as well as blood samples to examine changes in plasma levels of inflammatory markers, 5-HT, and tryptophan in order to look at possible underlying mechanisms of any changes seen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Major Depressive Disorder (MDD) by Mini International Neuropsychiatric Interview (MINI)
2. Current depressive episode with a MADRS score of ≥ 20
3. Males and females between ages 18 and 65
4. Able to understand and comply with the requirements of the study
5. Provision of written informed consent

Exclusion Criteria:

1. Use of any antidepressant drug
2. Use of any antibiotic drug in the past 4 weeks (may be eligible to participate after a 1-month washout period)
3. Use of any sleep medication in the past 4 weeks (may be eligible to participate after a 1-month washout period)
4. Milk, yeast, or soy allergy
5. History of alcohol or substance abuse in the past 6 months
6. Daily use of probiotic product in the past 2 weeks (may be eligible to participate after a 2-week washout period)
7. Use of any type of laxative
8. Consumption of products fortified in probiotics
9. Severely suicidal
10. Experiencing psychosis or bipolar episode
11. History of epilepsy or uncontrolled seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Mood | 8 weeks
  Mood will be assessed with the Montgomery-Asberg Depression Rating Scale (MADRS) with a cut-off score of 12 indicating remission.

SECONDARY OUTCOMES:
Anxiety | 8 weeks
  Anxiety will be assessed with the Generalized Anxiety Disorder Scale (GAD-7).
Cognition | 8 weeks
  Cognition will be assess with the Digit Symbol Substitution Test (DSST).
Sleep | 8 weeks
  Sleep will be assessed objectively using a polysomnogram to look at changes electrophysiological sleep architecture after 8 weeks of treatment.
Plasma | 8 weeks
  Plasma will be analyzed to look at levels of inflammatory markers to see whether there is a decrease after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, PhD, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Queen's University, Kingston, Ontario
  - Providence Care - Mental Health Services, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.